CLINICAL TRIAL: NCT04352127
Title: Comparison of Visual and Electromyography Assessments in Response to Train-of-Four Stimulation of the Ulnar Nerve
Brief Title: Visual and Electromyography Assessments in Response to Train-of-Four Stimulation of the Ulnar Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20-000619
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Neuromuscular Blockade; Tetragraph; AMG; EMG
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Dominant hand (Experimental): Subject scheduled to undergo an elective surgical procedure will have TetraGraph device lead placement on the dominant hand and routine clinical monitor on non-dominant hand
  Interventions: Device: TetraGraph
- Non-dominant hand (Experimental): Subject scheduled to undergo an elective surgical procedure will have TetraGraph device lead placement on the non-dominant hand and routine clinical monitor on dominant hand
  Interventions: Device: TetraGraph

INTERVENTIONS:
Device: TetraGraph — FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.

SUMMARY:
Researchers are comparing the accuracy of measuring muscle relaxation during and after surgery with a device that provides numeric value versus visual observation to count of muscle twitches or absence of them by a medical provider monitoring your anesthesia during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old
* Patients willing to participate and provide an informed consent
* Patients undergoing an elective surgical procedure that requires use of NMBA agents administered intraoperatively.

Exclusion Criteria:

* Patients with disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture, or any similar wrist injury.
* Patients with systemic neuromuscular diseases such as myasthenia gravis
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents, i.e., severe renal impairment or end-stage liver disease.
* Patients having surgery that would involve prepping the arm or leg into the sterile field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Dominant Hand: Subjects underwent an elective surgical procedure and had a TetraGraph device lead placement on the dominant hand and routine clinical monitor on non-dominant hand
  TetraGraph: FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.
- Non-dominant Hand: Subjects underwent an elective surgical procedure and had a TetraGraph device lead placement on the non-dominant hand and routine clinical monitor on dominant hand
  TetraGraph: FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.
Period: Overall Study
Arm/Group | Dominant Hand | Non-dominant Hand
Started | 29 | 26
Completed | 25 | 25
Not Completed | 4 | 1
Not completed — Unable to obtain readings | 4 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics was not collected for the Anesthesia providers
Groups:
- Total: Total of all reporting groups
Arm/Group | Dominant Hand | Non-dominant Hand | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Baseline characteristics were not collected for the Anesthesia providers
  years | 57.9 (13.1) | 57.9 (16.2) | 57.9 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics were not collected for the Anesthesia providers
  Participants
    Female | 16 | 17 | 33
    Male | 9 | 8 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Subjective Evaluation to Neurostimulation
Description: The percentage of subjective evaluations that overestimated the response of the adductor pollicis muscle following neurostimulation of the ulnar nerve when compared to objective measurements.
Time Frame: up to 1 hour postoperatively
Measure: Number; unit: percentage of evaluations
Arm/Group | Dominant Hand | Non-dominant Hand
Number analyzed (Participants) | 25 | 25
percentage of evaluations | 48.2 | 44.8

2. Secondary Outcome: Incidence of Residual Neuromuscular Blockade
Description: Number of subjects with train of four ratio < 0.9 after administration of reversal agent.
Time Frame: Up to 1 hour postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Dominant Hand | Non-dominant Hand
Number analyzed (Participants) | 25 | 25
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events will be collected from baseline to end of study, approximately 1 hour
Arm/Group | Dominant Hand | Non-dominant Hand
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT04352127/Prot_SAP_000.pdf